CLINICAL TRIAL: NCT03353948
Title: The Effect of Liraglutide on Pregnancy Rates in Obese Women With PCOS Undergoing in Vitro Fertilization: a Pilot Randomized Study
Brief Title: The Effect of a Liraglutide on IVF in Obese PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Vesna Salamun, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Obese PCOS IVF
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Polycystic Ovary Syndrome; Obesity; Infertility, Female
Keywords: Polycystic Ovary Syndrome; Obesity; Infertility; IVF
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity; Infertility, Female; Infertility | interventions — Liraglutide; Solutions; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metfrormin group (MET) (Active Comparator): Drug: Metformin
  Interventions: Drug: MET
- COMBI group (COMBI) (Active Comparator): Drug: liraglutide
  Interventions: Drug: COMBI

INTERVENTIONS:
Drug: MET — In the MET group metformin was initiated at a dose of 500 mg once per day and increased by 500 mg every 3 days up to 1000 mg BID per os for 12 weeks. After 1 month IVF was done.
  Other Names: Glucophage tbl
  Arms: Metfrormin group (MET)
Drug: COMBI — In the COMBI group the initial dose of MET was 500 mg for at least 2 wk and gradually increased to a final dose of 1000 mg BID. Liraglutide 1.2 mg QD s.c. was added after first two weeks of monotherapy with MET. After 1 month IVF was done.
  Other Names: Victoza 6 mg/ml solution for injection in pre-filled pen
  Arms: COMBI group (COMBI)

SUMMARY:
The aim of this study was to evaluate the impact of low dose liraglutide in combination with metformin compared to metformin alone on IVF pregnancy rate (PR) and cumulatively PR (IVF and spontaneous) in infertile obese women with PCOS who had been previously poor responders regarding weight reduction with lifestyle modification and resistant to first line reproductive treatments.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is the most common cause of anovulatory infertility, in particular when PCOS is linked to obesity. Obese PCOS has poor IVF outcomes associated with impaired oocyte and embryo parameters and morphology. The purpose of this pilot prospective study was to investigate the effect of the novel medical therapy (combination of metformin and liraglutide (COMBI)) in the specific infertile obese PCOS population. GLP-1 has been investigated in regulation of reproductive system in animal models. Current observations suggest that it directly regulates kisspeptin and GnRH expression and that ovaries express GLP-1 mRNA. In obese PCOS, GLP-1 receptor agonist liraglutide provided positive effects on weight reduction and glucose homeostasis

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to 38 years old
* polycystic ovary syndrome (rotterdam criteria)
* BMI of 30 kg/m² or higher
* Infertility
* Before IVF

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus

  * history of carcinoma
  * Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
  * personal or family history of MEN 2
  * significant cardiovascular, kidney or hepatic disease
  * the use of medications known or suspected to affect reproductive or metabolic functions
  * the use of statins, within 90 days prior to study entry no other ovarian pathology normal male semen

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
IVF pregnancy rates | 14 days
  Clinical pregnancy rate defined as the presence of a fetal heart beat by ultrasound
BMI | Patient's BMI was measured at the beginning and every four weeks during 12 weeks of clinical trial. ]
  Patient's BMI was defined as the patient's body mass in kilograms divided by the square of their height in meters.
Cumulative pregnancy rates | The pregnancies were collected by phone interview after one year
  Number of all pregnancies (IVF pregnancies and spontaneous pregnancies) per patient

SECONDARY OUTCOMES:
Oocyte nuclear maturation | 2 days
  The number of metaphase 2 oocytes, metaphase 1 oocytes, and germinal vesicles
Embryo quality | 6 days
  The embryo quality assessed by standard cleavage stage embryo grading system on day 3 of embryo culture. For any embryos grown to day 5, the embryo quality assessed by standard blastocyst grading system on day 5 of embryo culture

OTHER OUTCOMES:
The other outcomes was changes changes in fasting concentrations of glucose | Patient's fasting blood was drawn at the beginning and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Concentrations of fasting glucose was measured in mmol/L.
The other outcomes was changes changes in fasting concentrations of insulin | Patient's fasting blood was drawn at the beginning and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Fasting concentrations of insulin was measured in mU/L.
Other outcome was change in blood concentration of testosterone | Patient's fasting blood was drawn at the beginning and every four weeks during the 12 weeks of clinical trial. ]
  Patient's blood was drawn between 8 and 9 a.m. Blood concentration was measured in nmol/L.
Other outcome was change in blood concentration in androstenedione. | Patient's fasting blood was drawn at the beginning and every four weeks during the 12 weeks of clinical trial.
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of androstenedione was measured in nmol/L.
Other outcome was change in blood concentrations of SHBG (sex hormone-binding globulin). | Patient's fasting blood was drawn at the beginning and every four weeks during the 12 weeks of clinical trial. ]
  Patient's blood was drawn between 8 and 9 a.m. Blood concentrations of SHBG was measured in nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Vrtacnik Bokal, professor, Study Chair — UMC Ljubljana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jensterle Sever M, Kocjan T, Pfeifer M, Kravos NA, Janez A. Short-term combined treatment with liraglutide and metformin leads to significant weight loss in obese women with polycystic ovary syndrome and previous poor response to metformin. Eur J Endocrinol. 2014 Feb 7;170(3):451-9. doi: 10.1530/EJE-13-0797. Print 2014 Mar. PMID 24362411
- [Derived] Salamun V, Rizzo M, Lovrecic L, Hocevar K, Papler Burnik T, Janez A, Jensterle M, Vrtacnik Bokal E, Peterlin B, Maver A. The Endometrial Transcriptome of Metabolic and Inflammatory Pathways During the Window of Implantation Is Deranged in Infertile Obese Polycystic Ovarian Syndrome Women. Metab Syndr Relat Disord. 2022 Sep;20(7):384-394. doi: 10.1089/met.2021.0149. Epub 2022 Jul 13. PMID 35834645